CLINICAL TRIAL: NCT02973438
Title: Effects of Acute Intermittent Hypoxia (AIH) on Metabolism and Dysglycemia, in Overweight/Obese Persons With Spinal Cord Injuries (SCI)
Brief Title: Effects of Intermittent Hypoxia (IH) on Metabolism and Dysglycemia, in Overweight/Obese Persons SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20160818
Record Dates: First submitted 2016-11-18; First posted 2016-11-25 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injuries; Obesity; Insulin Resistance
Keywords: Spinal Cord Injuries; Obesity; Insulin Resistance; Intermittent hypoxia
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spinal Cord Injury (SCI) Intermittent Hypoxia then SHAM (Experimental): This arm of individuals with SCI will receive Intermittent Hypoxia (IH) and following a 3 week washout, SHAM treatment interventions.
  Interventions: Device: Intermittent Hypoxia (IH); Device: SHAM
- Control (CON) Intermittent Hypoxia then SHAM (Experimental): This arm of non injured control subjects will receive Intermittent Hypoxia (IH) and following a 3 week washout, SHAM treatment interventions.
  Interventions: Device: Intermittent Hypoxia (IH); Device: SHAM
- Spinal Cord Injury (SCI) SHAM then Intermittent Hypoxia (Experimental): This arm of individuals with SCI will receive SHAM and following a 3 week washout, Intermittent Hypoxia (IH) treatment interventions.
  Interventions: Device: Intermittent Hypoxia (IH); Device: SHAM
- Control (CON) SHAM then Intermittent Hypoxia (Experimental): This arm of non injured control subjects will receive SHAM and following a 3 week washout, Intermittent Hypoxia (IH) treatment interventions.
  Interventions: Device: Intermittent Hypoxia (IH); Device: SHAM

INTERVENTIONS:
Device: Intermittent Hypoxia (IH) — Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute hypoxic intervals (FIO2 = 0.09-0.12) with 3-minute normoxic intervals (FIO2 = 0.21). During hypoxic intervals, oxygen concentration may be adjusted to maintain participants SpO2 levels between 75-90%.
  Other Names: Hypoxico
Device: SHAM — Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute normoxic intervals (FIO2 = 0.21) with 3-minute normoxic intervals (FIO2 = 0.21).

SUMMARY:
The purpose of this research is to examine changes in blood glucose control and metabolism in individuals with SCI and non injured controls at rest and during exercise after five days of exposure to IH. This response will be compared with breathing normal room air (a SHAM control).

ELIGIBILITY:
Inclusion Criteria:

SCI only:

1. Lower extremity weakness or paralysis at C5 or below resulting from spinal cord injury for at least one year.
2. ASIA Classification A-D Overweight or obese as classified by a Body Mass Index (BMI) (kg/m2) of ≥ 25.0 (CON) and ≥ 22.0 (SCI).

SCI and non injured control:

Resting SaO2 ≥ 95%

Exclusion Criteria (SCI and non injured control):

1. Currently hospitalized
2. Resting heart rate ≥120 BPM
3. Resting systolic blood pressure >180 mm Hg
4. Resting diastolic Blood Pressure >100 mmHg
5. Self-reported history of unstable angina or myocardial infarction within the previous month
6. Previous cardiac surgery or condition that evidences ischemic heart disease
7. Cardiopulmonary complication such as COPD
8. Pregnancy determined by urine testing in sexually active females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Treatment Session (4 Days)
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia Then SHAM | Control (CON) Intermittent Hypoxia Then SHAM | Spinal Cord Injury (SCI) SHAM Then Intermittent Hypoxia | Control (CON) SHAM Then Intermittent Hypoxia
Started | 2 | 1 | 2 | 1
Completed | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Washout (Three Weeks)
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia Then SHAM | Control (CON) Intermittent Hypoxia Then SHAM | Spinal Cord Injury (SCI) SHAM Then Intermittent Hypoxia | Control (CON) SHAM Then Intermittent Hypoxia
Started | 2 | 1 | 2 | 1
Completed | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Second Treatment Session (4 Days)
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia Then SHAM | Control (CON) Intermittent Hypoxia Then SHAM | Spinal Cord Injury (SCI) SHAM Then Intermittent Hypoxia | Control (CON) SHAM Then Intermittent Hypoxia
Started | 2 | 1 | 2 | 1
Completed | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia Then SHAM | Control (CON) Intermittent Hypoxia Then SHAM | Spinal Cord Injury (SCI) SHAM Then Intermittent Hypoxia | Control (CON) SHAM Then Intermittent Hypoxia | Total
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 1 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 2
  Male | 2 | 0 | 2 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native Hawaiian | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardioendocrine Risk by Surrogate Blood Measures of the Homeostasis Model Assessment - Insulin Resistance (HOMA 2-IR)
Description: Insulin resistance was estimated by the Homeostasis Model Assessment of Insulin Resistance (HOMA2-IR), which is based on fasting glucose and insulin measurements. Values of > 1.8 were considered insulin resistant.
Time Frame: Baseline, day 5
Population: Unable to obtain blood samples from 2 participants in the control group and 1 participant withdrew prior to the baseline laboratory trial and therefore did not receive any intervention, therefore there is no reported data for the control group.
Measure: Mean (Standard Deviation); unit: IR Score
Groups:
- Spinal Cord Injury (SCI) Intermittent Hypoxia: This arm of individuals with SCI will receive Intermittent Hypoxia (IH). Intermittent Hypoxia (IH): Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute hypoxic intervals (FIO2 = 0.09-0.12) with 3-minute normoxic intervals (FIO2 = 0.21). During hypoxic intervals, oxygen concentration may be adjusted to maintain participants SpO2 levels between 75-90%.
- Control (CON) Intermittent Hypoxia: This arm of non injured control subjects will receive Intermittent Hypoxia (IH).
  Intermittent Hypoxia (IH): Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute hypoxic intervals (FIO2 = 0.09-0.12) with 3-minute normoxic intervals (FIO2 = 0.21). During hypoxic intervals, oxygen concentration may be adjusted to maintain participants SpO2 levels between 75-90%.
- Spinal Cord Injury (SCI) SHAM: This arm of individuals with SCI will receive SHAM. SHAM: Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute normoxic intervals (FIO2 = 0.21) with 3-minute normoxic intervals (FIO2 = 0.21).
- Control (CON) SHAM: This arm of non injured control subjects will receive SHAM. SHAM: Administered over a period of 5 consecutive days involving daily, hour long sessions of alternating 6-minute normoxic intervals (FIO2 = 0.21) with 3-minute normoxic intervals (FIO2 = 0.21).
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia | Control (CON) Intermittent Hypoxia | Spinal Cord Injury (SCI) SHAM | Control (CON) SHAM
Number analyzed (Participants) | 2 | 0 | 2 | 0
IR Score | 1.67 (0.91) |  | 1.60 (1.27) |

2. Secondary Outcome: Change in Exercise Substrate Partitioning as Measured Via VO2 Peak Test
Description: Change in exercise substrate partitioning as measured via endurance-maximal oxygen consumption (VO2peak test) and will be reported as change in carbohydrate oxidation (% of total energy expenditure).
Time Frame: Baseline, day 5
Measure: Mean (Standard Deviation); unit: % of total energy expenditure.
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia | Control (CON) Intermittent Hypoxia | Spinal Cord Injury (SCI) SHAM | Control (CON) SHAM.
Number analyzed (Participants) | 2 | 1 | 2 | 1
% of total energy expenditure. | 63.2 (25.7) | 64.9 (8.4) | 51.4 (23.6) | 70.9 (3.8)

ADVERSE EVENTS:
Time Frame: 29 days
Description: This study only collected treatment-emergent adverse events.
Arm/Group | Spinal Cord Injury (SCI) Intermittent Hypoxia | Control (CON) Intermittent Hypoxia | Spinal Cord Injury (SCI) SHAM | Control (CON) SHAM.
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02973438/Prot_SAP_000.pdf